CLINICAL TRIAL: NCT01401556
Title: Comparing Strategies Targeting Osteoporosis to Prevent Recurrent Fractures: C-STOP# Randomized Trial
Brief Title: C-STOP Fracture Trial
Acronym: C-STOP#
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00018520
Record Dates: First submitted 2011-07-06; First posted 2011-07-25 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2020-07

CONDITIONS: Osteoporosis
Keywords: osteoporosis; fracture; treatment; guidelines; quality
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Case Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Manager Intervention (Experimental): Osteoporosis case-managers will identify older fracture patients in Emergency Departments and Fracture Clinics; arrange bone mineral density (BMD) tests; meet with patients to counsel them and go over their results; and then offer and prescribe bisphosphonate treatment to those with low BMD.
  Interventions: Other: case management
- Multifaceted quality improvement intervention (Active Comparator): Active-comparator control consisting of telephone-based education for patients and treatment guidelines with reminders for family physicians
  Interventions: Other: Multifaceted quality improvement intervention

INTERVENTIONS:
Other: case management
  Arms: Case Manager Intervention
Other: Multifaceted quality improvement intervention
  Arms: Multifaceted quality improvement intervention

SUMMARY:
The objective of the proposed research is to improve quality of care for older outpatients who present to Emergency Departments and Fracture Clinics with an osteoporosis-related wrist or other upper extremity fracture. Although most of these patients warrant evidence-based and guideline-recommended osteoporosis testing and treatment, numerous studies demonstrate treatment rates less than 10-20% in the year post-fracture. Several trials, including the investigators own prior studies, have tried to address this osteoporosis care-gap and have reported that various multifaceted interventions (combinations of patient and physician education, guidelines, and physician reminders) can modestly improve treatment rates compared with usual care, although 60-70% of the patients exposed to these interventions still remain untreated. The investigators believe that a case-manager (who identifies and independently sees patients in clinic, arranges bone mineral density [BMD] tests, and offers guideline-based treatment to those with low BMD) represents a potential solution that holds great promise.

The investigators hypothesize that an osteoporosis case-manager will effectively and efficiently increase rates of osteoporosis treatment in older outpatients with upper extremity fractures when compared with a documented effective and cost-saving multifaceted intervention. To test this hypothesis the investigators propose a pragmatic patient-level randomized controlled comparative effectiveness trial with blinded outcomes ascertainment that compares the case-manager strategy with the multifaceted intervention.

DETAILED DESCRIPTION:
Objective: To improve treatment of osteoporosis in older patients with upper extremity fractures.

Background: Osteoporosis causes low bone mass and skeletal fragility leading to fractures of the hip, spine, and upper extremity that cause pain, deformity, disability, and even death. It affects 2 million older Canadians and costs us a billion dollars a year. Guidelines recommend aggressive treatment in older patients with osteoporosis-related fractures because risk of another fracture is 20% within 1-year and because bisphosphonate treatment reduces fracture risk by 50%. Unfortunately, less than 10% of older outpatients are treated for osteoporosis in the year post-fracture and even the most effective multifaceted interventions tested so far (i.e., combinations of patient education with physician guidelines and reminders) have only increased post-fracture osteoporosis treatment rates with bisphosphonates to 22%.

Proposed Strategy: Osteoporosis case-managers will identify older fracture patients in Emergency Departments and Fracture Clinics; arrange bone mineral density (BMD) tests; meet with patients to counsel them and go over their results; and then offer and prescribe bisphosphonate treatment to those with low BMD.

Hypothesis: An osteoporosis case-manager will effectively and efficiently increase rates of BMD testing and bisphosphonate treatment in older high-risk patients with upper extremity fractures compared with a previously tested effective and cost-saving multifaceted osteoporosis intervention (an active-comparator control consisting of telephone-based education for patients and treatment guidelines with reminders for family physicians).

Specific Aims: To determine whether an osteoporosis case-manager strategy can:

1. Increase rates of osteoporosis treatment more than a multifaceted intervention
2. Increase rates of BMD testing more than a multifaceted intervention
3. Be cost-effective when compared with either multifaceted intervention or usual care

Study Design: Randomized controlled comparative effectiveness trial with blinded (allocation-concealed) ascertainment of outcomes comparing case-managers to the multifaceted intervention. Eligible patients will be 50 years and older with an upper extremity fracture and not already treated with bisphosphonates, recruited from Emergency Departments and Fracture Clinics. Primary outcome will be the proportion starting bisphosphonates within 6-months. Secondary outcomes include BMD testing, any osteoporosis treatment, and appropriate care. Case-managers are expected to increase bisphosphonate treatment rates to 43% (achieved in our pilot trial) vs published multifaceted intervention rates of 22%. With alpha=0.05, beta=0.9, and 10% attrition rates, the total minimum required sample size is 240 patients. Using 1-year outcomes and micro-costing data from the trial and our published Markov decision analytic model for osteoporosis quality improvement interventions, the incremental costs and effectiveness of the case-manager will then be compared to both the multifaceted intervention and usual care. Major secondary outcome includes long-term treatment persistence, and to examine this question (e.g., 80% persistence rates with case-manager vs 50% persistence with multifaceted intervention) will require a sample size of at least 360 patients.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years or greater
* any forearm (distal radius or ulna, "wrist") or arm (proximal humerus, "upper arm") fracture

Exclusion Criteria:

* unable to give simple informed consent or unwilling to participate in the study
* unable to understand, read, and converse in English
* presence of pathological (e.g., cancer related) or multiple (e.g., major trauma) fractures
* already treated for osteoporosis with a bisphosphonate
* residence in a nursing home or from outside Edmonton

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Proportion of untreated patients newly starting prescription osteoporosis treatment with a bisphosphonate after their fracture | 6-months
  Proportion of previously untreated patients (%) newly starting prescription osteoporosis treatment with a bisphosphonate within 6-months of an upper extremity fragility fracture

SECONDARY OUTCOMES:
New Treatment Persistence | 1-year
  Of those newly starting treatment, what proportion are still persisting with it at 1-year of followup

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R Majumdar, MD, MPH, Principal Investigator — University of Alberta; Carrie Ye, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospitals, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Majumdar SR, Johnson JA, Bellerose D, McAlister FA, Russell AS, Hanley DA, Garg S, Lier DA, Maksymowych WP, Morrish DW, Rowe BH. Nurse case-manager vs multifaceted intervention to improve quality of osteoporosis care after wrist fracture: randomized controlled pilot study. Osteoporos Int. 2011 Jan;22(1):223-30. doi: 10.1007/s00198-010-1212-7. Epub 2010 Apr 1. PMID 20358359
- [Background] Majumdar SR, Johnson JA, McAlister FA, Bellerose D, Russell AS, Hanley DA, Morrish DW, Maksymowych WP, Rowe BH. Multifaceted intervention to improve diagnosis and treatment of osteoporosis in patients with recent wrist fracture: a randomized controlled trial. CMAJ. 2008 Feb 26;178(5):569-75. doi: 10.1503/cmaj.070981. PMID 18299546
- [Derived] McAlister FA, Ye C, Beaupre LA, Rowe BH, Johnson JA, Bellerose D, Hassan I, Majumdar SR. Adherence to osteoporosis therapy after an upper extremity fracture: a pre-specified substudy of the C-STOP randomized controlled trial. Osteoporos Int. 2019 Jan;30(1):127-134. doi: 10.1007/s00198-018-4702-7. Epub 2018 Sep 19. PMID 30232538